CLINICAL TRIAL: NCT07275879
Title: Evaluation of Quality of Life in Patients After Placement of a Modified Double J Ureteral Stent. Randomized Clinical Trial.
Brief Title: Evaluation of Quality of Life in Patients After Placement of a Modified Double J Ureteral Stent
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Luke's Clinical Hospital, Russia (Other)
Responsible Party: Principal Investigator, Mikheev Yury, Urologist, St. Luke's Clinical Hospital, Russia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21/4
Record Dates: First submitted 2025-11-18; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Ureteral Double-J Stent; Urolithiasis; Quality of Life
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (DJ stent) (Active Comparator): Non-prestented patients who will insert a standard DJ stent after surgery
  Interventions: Procedure: Ureteric stent insertion
- Group II (modified DJ stent) (Experimental): Non-prestented patients who will insert a modified DJ stent after surgery
  Interventions: Procedure: Ureteric stent insertion

INTERVENTIONS:
Procedure: Ureteric stent insertion — Ureteric stent insertion is the procedure to place a thin, flexible plastic tube that is temporarily in the ureter to help urine drain. They are placed with cystoscopic and X-ray guidances in an operating room setting

SUMMARY:
Double-J (DJ) stents are commonly inserted after ureteroscopy. There are several complications associated with the presence of DJ stent: urinary tract infection, stent encrustation, stent migration, and stent-related symptoms (SRS).

SRS occur in up to 80% of patients and include pain, hematuria, and dysuria, all of which negatively impact the patient's quality of life.

Physicians proposed the distal end of the ureteral stents might involve in SRS by over-simulating the trigone of bladder. The design of the distal end, made with a thinner loop than that of a standard DJ stent, is intended to mitigate SRS and reduce urine reflux.

DETAILED DESCRIPTION:
Study Design:

Prospective, randomized, open-label, controlled trial with two parallel arms.

Study Center:

Department of Urology, St. Luke's Clinical Hospital, St. Petersburg, Russia

Study Population:

All patients should not be prestented and should have no ureteral obstruction. 40 patients, divided into four equal groups of 20 people each:

Group I (standard DJ stent):

Group II (modified DJ stent)

Procedure for evaluation:

After surgery ( RIRS, ureteroscopy) reflux is assessed (gravity-filling cystogram). After stenting, the presence of post-stent reflux is assessed.

In the postoperative period, patients complete the USSQ (1st day, 7th day and before stent removal).

Statistics method:

The results are presented as the median and interquartile range (IQR) for continuous variables, and as frequencies (n with percentage %) for categorical variables. Statistical comparisons of all primary and secondary outcome measures between different treatment groups were conducted using the Mann-Whitney U test for continuous data. Meanwhile, categorical variables were analyzed using either Pearson's chi-square (χ²) test or Fisher's exact test, where appropriate. Thenthreshold for statistical significance was established at 5%, implying that a p-value less than 0.05 (p < 0.05) was considered statistically significant for all tests performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older
* Patients with kidney stones
* Patients with ureteral stones

Exclusion Criteria:

* Congenital anomalies of the urinary tract
* Urinary tract infections
* Upper urinary tract obstruction
* Complicated ureteroscopy (e.g., ureteral perforation)
* Pregnancy
* Pre-stented patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-28 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
ureteral reflux | Intraoperative
  Injection of raradiopaque dye using gravity- filling cystogram followed by X-ray imaging. If contrast entered or not entered the ureter and kidney, ureteral reflux was considered positive or not, respectively.
Assessment the Ureteral Stent Symptom Questionnaire (USSQ) | Postoperative: 1st and 7th day, before stent removal
  Ureteral stent symptom questionnaire (USSQ) a psychometrically valid measure to evaluate symptoms and impact on quality of life of ureteral stents.
  USSQ contains 38 questions and 2 visual analog scales (VAS), allowing assessment of the severity of SRS and their impact on the patient's quality of life. The questions are grouped into 6 domains:
  Urinary symptoms Pain General health Work performance Sexual matters Additional problems For each domain, a score index is calculated as the sum of the points from all questions in that domain. The scale scores range from 1 to 10, with higher values indicating more severe SRS and lower quality of life.

SECONDARY OUTCOMES:
Patient's height | Preoperative
  The patient's height is measured in centimeters.
Patient's weight | Preoperative
  The patient's weight is measured in centimeters.
Body mass index (BMI) | Preoperative
  Body mass index (BMI) is a value derived from the mass (weight) and height of a person.
  BMI = kg/m2
Operative time | Intraoperative (measured from start to end of procedure)
  total operative time in minutes
Surgery | Preoperative
  Type of surgery: ureteroscopy or retrograde intrarenal surgery or stenting

CONTACTS AND LOCATIONS:
Locations (1):
- St. Luke's Clinical Hospital, Saint Petersburg, Outside U.S./Canada, Russia

IPD SHARING:
Plan to Share IPD: No
We are currently finalizing our data sharing policy. All required individual participant data underlying the reported results will be made available for regulatory purposes immediately upon request, and may be shared with researchers following publication after de-identification, contingent on submission of a methodologically sound proposal and compliance with institutional and national privacy regulations